CLINICAL TRIAL: NCT06605547
Title: The Effect of Injectable Platelet-Rich Fibrin As An Adjunct to Non-Surgical Periodontal Therapy on Clinical Parameters in Smokers With Periodontitis: A Split-Mouth Randomized Controlled Trial
Brief Title: The Effect of I-PRF As An Adjunct to Non-Surgical Periodontal Therapy on Clinical Parameters in Smokers With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Bilge MERACI YILDIRAN, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAIBU-SBF-BMY-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Periodontitis
Keywords: smoker; periodontitis; i-PRF
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Split-mouth, randomized controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): Test sites receiving the subgingival application of i-PRF after NSPT.
  Interventions: Procedure: Non-surgical periodontal treatment; Other: Subgingival application of i-PRF
- Control group (Placebo Comparator): Control sites treated with saline after NSPT.
  Interventions: Procedure: Non-surgical periodontal treatment; Device: Subgingival application of saline

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — The non-surgical periodontal treatment (scaling and root planing) was applied under local anesthesia using ultrasonic device and Gracey curettes. After scaling and root planing, periodontal pockets were irrigated using saline solution. Non-surgical periodontal treatment was completed in one or two sessions within 24 hours.
Device: Subgingival application of saline — For the subgingival saline application at the control sites, the insulin needle was filled with saline and the 29-gauge needle tip was gently placed into the periodontal pocket. The saline was injected into the periodontal pocket until it was seen to overflow from the gingival margin. Subgingival saline application was repeated on the 7th day.
  Arms: Control group
Other: Subgingival application of i-PRF — For subgingival application of i-PRF at the test sites, the i-PRF taken into the insulin syringe, the 29-gauge needle tip was gently placed into the periodontal pocket and the i-PRF was injected into the periodontal pocket until it reached the gingival margin (until it overflowed from the sulcus). Subgingival i-PRF application was repeated on the 7th day.
  Arms: Test group

SUMMARY:
The aim of this clinical trial is to evaluate the effect of subgingival injectable platelet-rich fibrin (i-PRF) application on clinical periodontal parameters as an adjunct to non-surgical periodontal treatment (NSPT) in smokers with periodontitis.

Twenty-five systemically healthy, smoker patients with stage II/III periodontitis were included in the study. In this split-mouth trial, subgingival i-PRF was applied to the test group in addition to NSPT, while saline was applied to the control group after NSPT. Subgingival i-PRF/saline application was repeated on the 7th day in both groups. Clinical periodontal parameters were recorded at baseline, 1st and 3rd months after the treatment.

DETAILED DESCRIPTION:
Twenty-five systemically healthy, smoker patients with periodontitis were included in the study. All individuals were examined at baseline, 1st and 3rd months after non-surgical periodontal treatment including, whole mouth probing pocket depth (PPD), clinical attachment loss (CAL), presence of bleeding on probing (BOP), gingival index (GI) and Turesky Modified Quigley-Hein Plaque Index (TQHPI) except the third molars. PPD and CAL were measured at six sites per tooth using a manual periodontal probe. All measurements and NSPT were performed by the same blinded and calibrated examiner (TCG).

The NSPT included supra- and subgingival scaling, root planing and oral hygiene instructions. Subgingival scaling and root planing were performed under local anesthesia within the 24 h. After NSPT, four contralateral deep pockets (two for each side) in premolar/molar ares were determined. The sites were randomly divided into test sites receiving the subgingival application of i-PRF and controls treated with saline.

After the NSPT was completed, the i-PRF was produced as follows: 9 mL of whole blood was collected from the antecubital vein in a sterile plastic tubes without anticoagulant and immediately centrifuged at 700 rpm for 3 minutes with a centrifuge device. After centrifugation, the upper liquid layer was collected as i-PRF and placed into an insulin syringe connected to a 29G needle.

Before the i-PRF application, the teeth were isolated with a cotton roll and dried with a cotton pellet. The 29-gauge needle tip was gently placed into the periodontal pocket and the i-PRF was injected into the periodontal pocket until it reached the gingival margin (until it overflowed from the sulcus). For the subgingival saline application, the insulin syringe was filled with saline and the 29-gauge needle tip was gently placed into the periodontal pocket. The saline was injected into the periodontal pocket until it was seen to overflow from the gingival margin. After the subgingival application of i-PRF/saline , the application areas were isolated and waited for 10 minutes in order to prevent the i-PRF from being removed from the sulcus with oral fluids until it turned into a gel. Subgingival i-PRF/salin application was performed by a periodontist (BMY).Patients were instructed not to drink or eat anything, including water, for at least 30 minutes after the procedure. Patients were informed about oral hygiene practices (tooth brushing and interdental cleaning) and were motivated to perform daily oral care. Patients were given an appointment for the second application of i-PRF/salin application 7 days later. In this session, i-PRF/salin application was applied to the previously applied areas, oral hygiene was checked and patients were informed again. Patients were called again in the 1st and 3rd months, periodontal clinical measurements were repeated and oral hygiene motivation was given.

Statistical analyses were performed using a statistical analysis software (SPSS v.25.0; IBM). The Shapiro Wilk test was used to determine the normality of the present data and the variance homogeneity was checked with the Levene test. For non-normally distributed data, the Mann Whitney U test was used for pairwise comparison. The Independent Samples T test was performed for normally distributed data. The Friedman test was used to examine the differences between three dependent groups. Bonferroni correction was performed for multiple variations. The statistical significance value was accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients were systemically healthy adults,
* having at least 20 natural teeth,
* the presence of contralateral periodontal pockets (PPD≥ 5 mm) and CAL≥2 mm on a minimum of two premolar/molar teeth on each side and no furcation involvement,
* smoking more than 10 cigarettes per day for at least 5 years,
* stage II-III periodontitis patients

Exclusion Criteria:

* individuals had past periodontal treatment within 6 months
* individuals had used systemic antibiotics in the last 6 months or anti- inflammatory drugs in the last 3 months before the beginning of the trial,
* patient with clotting and hematologic disorders, had used drugs affecting the natural coagulation process,
* patients taking medications that affect the gingival and periodontal tissues
* pregnant or breastfeeding females

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | Baseline, 1st and 3rd months
  CAL measured as the change in distance from the cementoenamel junction to the bottom of the gingival sulcus (the most coronal attachment) using a Williams periodontal probe. The changes in clinical attachment loss was measured for determining the severity of disease.
Probing pocket depth (PPD) | Baseline, 1st and 3rd months
  PPD measured as the change in distance from the gingival margin to the bottom of the gingival sulcus using a Williams periodontal probe. The changes in PPD was measured for determining of the severity of disease and clinical outcome.

SECONDARY OUTCOMES:
Bleeding on probing (BOP) | Baseline, 1st and 3rd months
  All six sites of all teeth were probed to assess whether this elicited bleeding (+) or not (-). The severity of gingival inflammation was expressed as a percentage (BOP=number of bleeding sites×100/number of sites evaluated). Bleeding on probing was recorded for classifying and evaluating gingival inflammation
Turesky Modified Quigley-Hein Plaque Index (TQHPI) | Baseline, 1st and 3rd months
  TQHPI for the entire mouth was determined by dividing the total score by the number of surfaces examined. Scoring was as follows:
  * 0: no plaque
  * 1: separate flecks of plaque at the cervical margin of the tooth
  * 2: a thin continuous band of plaque (≤ 1 mm) at the cervical margin of the tooth
  * 3: a band of plaque > 1 mm but covering less than one-third of the crown of the tooth
  * 4: plaque covering at least one-third but less than two- thirds of the crown of the tooth
  * 5: plaque covering two-thirds or more of the crown of the tooth labial/buccal and lingual surfaces assessed after using a disclosing solution.
  TQHPI was recorded for determining and classifying oral hygiene status.
Gingival index (GI) | Baseline, 1st and 3rd months
  To determine the gingival index (Löe & Silness), gingival bleeding caused by running a Williams periodontal probe inside the pocket on the mesial, distal, buccal, and palatal surfaces of all teeth was evaluated. The gingival index of an individual was obtained by summing the values determined for each tooth and calculating the averages. Scoring was as follows:
  * 0: Healthy gums.
  * 1: Mild discolouration and oedematous gingiva. No bleeding on probing.
  * 2: Red, oedematous and shiny gingiva. There is bleeding on probing.
  * 3: Red, oedematous and ulcerated gingiva. There is spontaneous bleeding. Gingival index was recorded for classifying and evaluating sulcular gingival inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cagiran Gurbuz T, Meraci Yildiran B. The clinical efficacy of injectable platelet-rich fibrin (i-PRF) as an adjunct to nonsurgical periodontal therapy in smokers with periodontitis. BMC Oral Health. 2025 Apr 23;25(1):618. doi: 10.1186/s12903-025-06019-w. PMID 40269777